CLINICAL TRIAL: NCT01732809
Title: Fields of Effects of Two Commercial Preparations of Botulinum Toxin Type A at Equal Labeled Unit Doses
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hexsel Dermatology Clinic (Other)
Responsible Party: Principal Investigator, Doris Hexsel, MD, Hexsel Dermatology Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 11-2011
Record Dates: First submitted 2012-11-07; First posted 2012-11-26 (Estimated); Results first posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-11

CONDITIONS: Skin Wrinkling
Keywords: wrinkles; botulinum toxin; abobotulinumtoxinA; onabotulinumtoxinA; field of anhydrotic effects
MeSH Terms: interventions — abobotulinumtoxinA; Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- abobotulinumtoxin A (Active Comparator): Patients were randomized to the side of the forehead (left or right) in which the products were administered. All the patients received abobotulinumtoxin A in one of the sides of the forehead.
  Interventions: Drug: AbobotulinumtoxinA (ABO)
- onabotulinumtoxin A (Active Comparator): Patients were randomized to the side of the forehead (left or right) in which the products were administered. All the patients received onabotulinumtoxin A in one of the sides of the forehead.
  Interventions: Drug: OnabotulinumtoxinA (ONA)

INTERVENTIONS:
Drug: AbobotulinumtoxinA (ABO) — Isovolumetric (0.02 mL) doses of 2 units of abobotulinumtoxinA injected on one side of the forehead.
  Other Names: Dysport®
  Arms: abobotulinumtoxin A
Drug: OnabotulinumtoxinA (ONA) — Isovolumetric (0.02 mL) doses of 2 units of onabotulinumtoxinA injected on the other side of the forehead.
  Other Names: Botox®
  Arms: onabotulinumtoxin A

SUMMARY:
The purpose of this study is to assess the fields of anhydrotic effect (FAE) of abobotulinumtoxinA and onabotulinumtoxinA at the same labeled unit dose (1:1 units), comparing both sweat gland and muscle activity.

DETAILED DESCRIPTION:
This is a prospective, single-center, randomized, double-blind study. All participants were recruited from a research center in Porto Alegre, Brazil, and provided written informed consent. The purpose of this study is to assess the fields of anhydrotic effect (FAE) of abobotulinumtoxinA and onabotulinumtoxinA at the same labeled unit dose (1:1 units), comparing both sweat gland and muscle activities. Nineteen patients were enrolled and evaluations were performed at baseline and 28 days after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Signed consent
2. Female subjects aged between 18 to 60 years
3. Phototype I to IV
4. Moderate to severe wrinkles in the forehead region on maximal contracture of the frontalis muscle according to the Wrinkle Severity Scale
5. Subjects with the Minor Test* considered positive from grade 3 to 5 on the Minor test sweat intensity scale, showing sweat on the forehead under standardized conditions
6. Medical history and clinical examination that, in the investigator's opinion, do not prevent the subject from participating in the study or from using the proposed medication
7. Negative urinary pregnancy test at the initial visit for women of childbearing potential
8. Use of an effective contraceptive method (oral or injectable contraception, abstinence, intrauterine device, diaphragm, hysterectomy or bilateral ovariectomy, tubal attachment, condom, sponge, spermicide or partner with vasectomy) throughout the study for women of childbearing potential
9. Subjects must agree not to undergo other dermatological or aesthetic treatments during the study period *The Minor test must be the last test to be done. Only the subjects who fulfill all the inclusion criteria above undergo the Minor test to check for sweating in the frontal region. The graduation considered positive for inclusion in the study will be 3 to 5.

Inclusion Criteria:

1. Pregnancy or intention to become pregnant during the study period
2. Breastfeeding
3. Botulinum toxin treatments in the last 6 months
4. Subjects participating in other clinical studies
5. Any surgical procedure performed that has affected the frontal or orbicularis muscle, previous blepharoplasty or eyebrow raising
6. Any cosmetic procedures, including fillers, or scars that may interfere with the results of the study
7. Fronto-parietal alopecia according to the Norwood-Hamilton classification
8. Neoplastic, muscular or neurological diseases
9. Use of using aminoglycoside antibiotics or penicillamines, quinine or calcium channel blockers or that they will use at any time during the study
10. Inflammatory or infectious processes at the application site
11. Evident facial asymmetry
12. History of adverse event, such as sensitivity to the components of the formula, ptosis or any other adverse event that, in the investigator's opinion, prevents the research subject from participating in the study
13. Myasthenia Gravis, Eaton-Lambert Syndrome and motor neuron disease
14. Coagulation disorders or use of anticoagulants
15. Autoimmune disease
16. History of poor adherence to treatments or who have shown lack of cooperation to adhere to the study protocol
17. Any condition that, in the investigator's opinion, could compromise the results of the study

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2011-01; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Doris M Hexsel, MD, Principal Investigator — Brazilian Center for Studies in Dermatology
Locations (1):
- Brazilian Center for Studies in Dermatology, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Hexsel D, Hexsel C, Siega C, Schilling-Souza J, Rotta FT, Rodrigues TC. Fields of effects of 2 commercial preparations of botulinum toxin type A at equal labeled unit doses: a double-blind randomized trial. JAMA Dermatol. 2013 Dec;149(12):1386-91. doi: 10.1001/jamadermatol.2013.6440. PMID 24108521

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: sides of the forehead
Groups:
- Group A: Patients received 2U/0.02mL of reconstituted abobotulinumtoxinA on the right side of the forehead and 2U/0.02mL of reconstituted onabotulinumtoxinA on the left side.
- Group B: Patients received 2U/0.02mL of reconstituted abobotulinumtoxinA on the left side of the forehead and 2U/0.02mL of reconstituted onabotulinumtoxinA on the right side.
Period: Overall Study
Arm/Group | Group A | Group B
Started | 9; 18 sides of the forehead | 10; 20 sides of the forehead
Completed | 9; 18 sides of the forehead | 9; 18 sides of the forehead
Not Completed | 0; 0 sides of the forehead | 1; 2 sides of the forehead

BASELINE CHARACTERISTICS:
Population: Split-face study. Each patient was treated with abobotulinumtoxin A in one side of the forehead, and with onabotulinumtoxin A on the contralateral side. Sides were randomized.
Units Other Than Participants: Sides of the forehead
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 9 | 10 | 19
Number analyzed (Sides of the forehead) | 18 | 20 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.7 (10.6) | 35.7 (9.1) | 39.0 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 9 | 10 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Brazil | 9 | 10 | 19

OUTCOME MEASURES:

1. Primary Outcome: Horizontal Diameter of the Fields of Anhidrotic Effect
Description: The Horizontal Diameter of the Fields of Anhidrotic Effect were measured with Mirror Medical Imaging Software (Canfield Scientific, Inc., Parsippany, NJ)
  The injection of botulinum toxin type A causes both muscle paralysis and anhydrosis on sweat glands activity. The size of the muscular and anhydrotic effects are called field of anhidrotic effects (FAE) and field of muscular effects (FME). The reaction of iodine and starch with the sweat (Minor's test) allows visualizing the field of anhidrotic effects and measuring them.
  The peak effect of botulinum toxin type A occurs between 15 and 30 days after injection. There is no change from the baseline, because no FAE are observed at baseline.
Time Frame: 28 days
Population: Per protocol.
Measure: Mean (Standard Deviation); unit: centimeters
Groups:
- Abobotulinumtoxin A; Onabotulinumtoxin A: Patients were randomized to the side of the forehead (left or right) in which the products were administered.
Arm/Group | Abobotulinumtoxin A | Onabotulinumtoxin A
Number analyzed (Participants) | 18 | 18
centimeters | 0.84 (0.14) | 1.24 (0.24)

2. Primary Outcome: Vertical Diameter of the Fields of Anhidrotic Effect
Description: The Vertical Diameter of the Fields of Anhidrotic Effect were measured with Mirror Medical Imaging Software (Canfield Scientific, Inc., Parsippany, NJ)
  The injection of botulinum toxin type A causes both muscle paralysis and anhydrosis on sweat glands activity. The size of the muscular and anhydrotic effects are called field of anhidrotic effects (FAE) and field of muscular effects (FME). The reaction of iodine and starch with the sweat (Minor's test) allows visualizing the field of anhidrotic effects and measuring them.
  The peak effect of botulinum toxin type A occurs between 15 and 30 days after injection. There is no change from the baseline, because no FAE are observed at baseline.
Time Frame: 28 days
Population: Per protocol
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Abobotulinumtoxin A | Onabotulinumtoxin A
Number analyzed (Participants) | 18 | 18
centimeters | 1.19 (0.19) | 1.50 (0.26)

3. Primary Outcome: Area of the Fields of Anhidrotic Effect
Description: The area of the Fields of Anhidrotic Effect were measured with Mirror Medical Imaging Software (Canfield Scientific, Inc., Parsippany, NJ)
  The injection of botulinum toxin type A causes both muscle paralysis and anhydrosis on sweat glands activity. The size of the muscular and anhydrotic effects are called field of anhidrotic effects (FAE) and field of muscular effects (FME). The reaction of iodine and starch with the sweat (Minor's test) allows visualizing the field of anhidrotic effects and measuring them.
  The peak effect of botulinum toxin type A occurs between 15 and 30 days after injection. There is no change from the baseline, because no FAE are observed at baseline.
Time Frame: 28 days
Population: Per protocol.
Measure: Mean (Standard Deviation); unit: centimeters squared
Arm/Group | Abobotulinumtoxin A | Onabotulinumtoxin A
Number analyzed (Participants) | 18 | 18
centimeters squared | 0.86 (0.22) | 1.49 (0.49)

4. Secondary Outcome: Wrinkle Severity Scale (WSS) at Maximum Contraction
Description: It is a 4-point validated scale for forehead lines:
  0 - None
  1. - Mild
  2. - Moderate
  3. - Severe
  The injection of botulinum toxin type A causes both muscle paralysis and anhydrosis on sweat glands activity. The size of the muscular and anhydrotic effects are called field of anhidrotic effects (FAE) and field of muscular effects (FME). The muscular effect reduction can be observed by the reduction of facial lines.
  Wrinkle scales are used to grade the muscular effects of botulinum toxin.
  The peak effect of botulinum toxin type A occurs between 15 and 30 days after injection. There is no change from the baseline, because no FME are observed at baseline.
Time Frame: Baseline and 28 days
Population: Per protocol.
Measure: Number; unit: participants
Arm/Group | Abobotulinumtoxin A | Onabotulinumtoxin A
Number analyzed (Participants) | 18 | 18
participants
  Baseline - Grade 0 | 0 | 0
  Baseline - Grade 1 | 0 | 0
  Baseline - Grade 2 | 7 | 6
  Baseline - Grade 3 | 11 | 12
  At 28 days - Grade 0 | 5 | 6
  At 28 days - Grade 1 | 10 | 8
  At 28 days - Grade 2 | 2 | 3
  At 28 days - Grade 3 | 1 | 1

5. Secondary Outcome: Wrinkle Severity Scale (WSS) at Rest
Description: It its a 4-point validated scale for forehead lines:
  0 - None
  1. - Mild
  2. - Moderate
  3. - Severe
  The injection of botulinum toxin type A causes both muscle paralysis and anhydrosis on sweat glands activity. The size of the muscular and anhydrotic effects are called field of anhidrotic effects (FAE) and field of muscular effects (FME). The muscular effect reduction can be observed by the reduction of facial lines.
  Wrinkle scales are used to grade the muscular effects of botulinum toxin.
  The peak effect of botulinum toxin type A occurs between 15 and 30 days after injection. There is no change from the baseline, because no FME are observed at baseline.
Time Frame: Baseline and 28 days
Population: Per protocol.
Measure: Number; unit: participants
Arm/Group | Abobotulinumtoxin A | Onabotulinumtoxin A
Number analyzed (Participants) | 18 | 18
participants
  Baseline - Grade 0 | 1 | 1
  Baseline - Grade 1 | 8 | 7
  Baseline - Grade 2 | 4 | 5
  Baseline - Grade 3 | 5 | 5
  At 28 days - Grade 0 | 10 | 10
  At 28 days - Grade 1 | 6 | 6
  At 28 days - Grade 2 | 2 | 2
  At 28 days - Grade 3 | 0 | 0

6. Secondary Outcome: Evoked Compound Muscle Action Potentials (ECMAP)
Description: Amplitude of the evoked compound muscle action potentials in the frontalis muscle on stimulation of the facial nerve performed at baseline and visit 2 using surface electrodes on the forehead and electrical stimulation of the facial nerve according to standard neurophysiologic procedures.
  The amplitude of the ECMAP was performed by an experienced neurologist using an electromyography device (Teca Sapphire; Teca Corp).
Time Frame: Baseline and 28 days
Population: Per protocol.
Measure: Mean (Standard Deviation); unit: microvolts
Arm/Group | Abobotulinumtoxin A | Onabotulinumtoxin A
Number analyzed (Participants) | 18 | 18
microvolts
  Baseline | 1108.17 (364.76) | 1079.11 (266.02)
  Day 28 | 202.89 (258.44) | 165.39 (232.10)

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Abobotulinumtoxin A | Onabotulinumtoxin A
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 2/19 | 1/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abobotulinumtoxin A (N=19) | Onabotulinumtoxin A (N=19)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) — Erythema after injection procedure
Bleeding (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) — Minimal bleeding after injection procedure

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No